CLINICAL TRIAL: NCT04624178
Title: Phase II Study of Rucaparib and Nivolumab in Patients With Leiomyosarcoma
Brief Title: A Study of Rucaparib and Nivolumab in People With Leiomyosarcoma
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: Bristol-Myers Squibb (Industry); Clovis Oncology, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20-358
Record Dates: First submitted 2020-11-05; First posted 2020-11-10 (Actual); Last update posted 2025-11-20 (Actual); Status verified 2025-11

CONDITIONS: Leiomyosarcoma
Keywords: Rucaparib; Nivolumab; 20-358
MeSH Terms: conditions — Leiomyosarcoma | interventions — rucaparib; Nivolumab

STUDY DESIGN:
Intervention Model Description: This is a Phase II open label study evaluating the combination of rucaparib and nivolumab in patients with refractory LMS.
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Rucaparib in combination with Nivolumab (Experimental): One treatment cycle will consist of 28 days. Patients will receive rucaparib at 600 mg, orally, twice daily, continuously for 28 days. They will receive 480mg of nivolumab intravenously on day 1 of every four-week cycle. This is the recommended phase II dose of the combination therapy. Re-staging scans will be performed every 8 weeks.
  Treatment will be repeated until the patient develops progressive disease or unacceptable toxicity or for a maximum duration of 26 cycles as long as patients are receiving benefit from treatment, have not had disease progression, met any criteria for study withdrawal and are tolerating therapy.
  Interventions: Drug: Rucaparib; Drug: Nivolumab

INTERVENTIONS:
Drug: Rucaparib — Rucaparib at 600 mg, orally, twice daily, continuously for 28 days.
Drug: Nivolumab — Nivolumab 480mg intravenously on day 1 of every four-week cycle.

SUMMARY:
The purpose of this study is to find out whether combining the study drugs rucaparib and nivolumab may be an effective treatment for advanced and/or metastatic LMS, and whether the study treatment works as well as the standard chemotherapy for this type of cancer.

ELIGIBILITY:
Inclusion Criteria:

* Male or female age ≥ 18 years at the time of informed consent
* Be willing and able to provide written informed consent/assent for the trial
* Be willing to comply with treatment protocol
* Subjects must have a histologically confirmed unresectable/metastatic LMS
* Availability of archival tissue for correlative studies. Either a paraffin block or at least 20 unstained slides are acceptable
* Adequate performance status: ECOG 0 - 2
* Subjects must have had at least 1 but not more than 3 prior lines of systemic therapy (e.g. chemotherapy, immunotherapy, targeted or biological therapy) for their LMS. Patients who decline the standard of care first-line systemic therapy will be eligible for this trial. Prior adjuvant therapy will not count provided it was completed more than 6 months previously.
* Presence of measurable disease per RECIST v1.1. Target lesions must not be chosen from a previously irradiated field unless there has been radiographically and/or pathologically documented tumor progression in that lesion prior to enrollment.
* Adequate organ function determined within 14 days of treatment initiation, defined as per Hematological
* Absolute neutrophil count (ANC) ≥1.5 K/mcL
* Platelets ≥100 K/ mcL
* Hemoglobin ≥9 g/dL Renal
* Serum creatinine OR Measured or calculated creatinine clearance Estimated glomerular filtration rate (eGFR) ≥ 30 mL/min/1.73 m2. For calculated CrCL, the Cockcroft Gault formula or institutional standard formula can be used.

Hepatic

* Serum total bilirubin <1.5 X ULN OR <2 X ULN if hyperbilirubinemia is due to Gilbert's syndrome
* AST (SGOT) and ALT (SGPT) Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤ 3 × upper limit of normal (ULN); if liver metastases, then ≤ 5 × ULN Coagulation
* International Normalized Ratio ≤1.5 X ULN (≤ 2.5 × ULN if on anticoagulants)
* Women of childbearing potential must have a negative serum pregnancy test at screening and ≤ 72 hours prior to the first dose of study treatment.
* Female subjects of childbearing potential must be willing to use an adequate method of contraception as outlined in Section 15.1.6 and not breastfeed, for the duration of the study and for at least 6 months after the last after the last dose of study medication.

Note: Abstinence is acceptable if this is the usual lifestyle and preferred contraception for the subject.

* Non-sterile male subjects and their female partners must be willing to use a highly effective method of contraception during the study treatment period and for at least 7 months after the last dose of study treatment. Nonsterile males must avoid sperm donation for the duration of the study and for at least 7 months after last study drug.
* Patients who were treated with chemotherapy or any investigational therapies or other anti-cancer agent, if eligible, must have been completed at least 3 weeks or at least 5 half-lives (whichever is longer, but no less than 3 weeks) before the study drug administration. All AEs must be ≤ NCI CTCAE v5 Grade 1, except alopecia and stable neuropathy, which must have resolved to Grade ≤ 2 or baseline. Patients who were treated with estrogen modulating therapies (aromatase inhibitors, tamoxifen, GnRH agonists etc.) must have been treated at least 2 weeks prior to study drug administration.
* Patients who were treated with radiotherapy must have completed radiation therapy at least 2 weeks before the study drug administration.
* Must be willing to agree to an on-treatment biopsy if deemed safe and feasible by the treating physician

Exclusion Criteria:

* Uncontrolled intercurrent illness including current active or chronic infection requiring systemic therapy or the following cardiac criteria:

  * Symptomatic congestive heart failure (NYHA classification III or IV) within 6 months
  * Acute myocardial infarction ≤6 months prior to Day 1
  * Grade ≥2 ventricular arrhythmia ≤6 months prior to Day 1
  * History of cerebrovascular accident within 6 months before first dose of study drugs
* Has known active central nervous system (CNS) metastases and/or carcinomatous meningitis. Patients with previously treated brain metastases may participate provided they are stable (without evidence of progression by imaging for at least four weeks prior to the first dose of trial treatment and any neurologic symptoms have returned to baseline), have no evidence of new or enlarging brain metastases, and are not using steroids for at least 7 days prior to trial treatment. This exception does not include carcinomatous meningitis which is excluded regardless of clinical stability.
* Evidence of clinically significant immunosuppression such as the following:

  * Primary immunodeficiency state such as Severe Combined Immunodeficiency Disease
  * Concurrent opportunistic infection
  * Receiving systemic immunosuppressive therapy (> 2 weeks) including oral steroid doses > 10 mg/day of prednisone or equivalent within 7 days prior to enrollment. However, in the setting of non-immune mediated indications for steroid use, chronic/active low dose steroid use may be permitted at the discretion of the principal investigator. The dose of steroid allowed in this setting is also at the discretion of the principal investigator. (Use of inhaled or topical steroids is permitted.)
* History or evidence of symptomatic autoimmune disease (e.g., pneumonitis, glomerulonephritis, vasculitis, or other), or history of active autoimmune disease that has required systemic treatment (i.e., use of corticosteroids, immunosuppressive drugs or biological agents used for treatment of autoimmune diseases) in past 2 years prior to enrollment. Replacement therapy (e.g., thyroxine for hypothyroidism, insulin for diabetes or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency) is not considered a form of systemic treatment for autoimmune disease.
* Known history of a positive test for human immunodeficiency virus (HIV) or known acquired immunodeficiency syndrome (AIDS). Has known active Hepatitis B (e.g., HBsAg reactive) or Hepatitis C (e.g., HCV RNA [qualitative] is detected).
* History of non-viral hepatitis or cirrhosis
* A history of alcohol abuse
* Use of any live vaccines (e.g., against infectious diseases such as varicella) within 4 weeks (28 days) of initiation of study therapy
* Has a known history of active TB (Bacillus Tuberculosis)
* Prior therapy with a PARP inhibitor and/or PD-1/PD-L1 monoclonal antibody is not permitted.

  * Patients who have not recovered from clinically significant adverse events of prior therapy to ≤ NCI CTCAE v5 Grade 1, except alopecia and stable neuropathy, which must have resolved to Grade ≤ 2 or baseline. Except for AEs not considered a likely safety risk (e.g., alopecia, neuropathy)
  * Note: If subject received major surgery, they must have recovered adequately from the toxicity and/or complications from the intervention prior to starting therapy events due to a previously administered agent.
* Presence of a gastrointestinal condition that may affect drug absorption
* Known allergy or reaction to any component of either study drug formulation
* Has evidence of active, non-infectious pneumonitis.
* Women who are pregnant or breast feeding
* Subjects expecting to have a child within the projected duration of the trial, starting with the pre-screening or screening visit through 6 months after the last dose of study treatment(s) for women or 7 months for men.
* Presence of any other concurrent malignancy requiring active therapy or thought to potentially interfere with the safe conduct or assessment of outcomes on this trial
* Prior allogeneic stem cell transplantation or organ transplantation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2020-11-05 (Actual); Primary Completion 2026-11-16 (Estimated); Study Completion 2026-11-16 (Estimated)

PRIMARY OUTCOMES:
Best objective response rate | by 24 weeks
  as assessed by RECIST 1.1

SECONDARY OUTCOMES:
Progression free survival (PFS) | at 24 weeks
  PFS is defined as the period from start of study treatment until recurrent or progressive of disease (POD) is objectively documented (taking as reference for progressive disease the smallest measurement recorded on study), death, or date of last study visit involving assessment of disease status.

CONTACTS AND LOCATIONS:
Overall Officials: Sujana Movva, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (7):
- United States (7):
  - Memorial Sloan Kettering Basking Ridge (Limited Protocol Activities), Basking Ridge, New Jersey
  - Memorial Sloan Kettering Monmouth (Limited Protocol Activities), Middletown, New Jersey
  - Memorial Sloan Kettering Bergen (Limited Protocol Activities), Montvale, New Jersey
  - Memorial Sloan Kettering Commack (Limited protocol activities), Commack, New York
  - Memorial Sloan Kettering Westchester (Limited Protocol Activities), Harrison, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Memorial Sloan Kettering Nassau (Limited Protocol Activities), Uniondale, New York

IPD SHARING:
Plan to Share IPD: Yes
Memorial Sloan Kettering Cancer Center supports the international committee of medical journal editors (ICMJE) and the ethical obligation of responsible sharing of data from clinical trials. The protocol summary, a statistical summary, and informed consent form will be made available on clinicaltrials.gov when required as a condition of Federal awards, other agreements supporting the research and/or as otherwise required. Requests for deidentified individual participant data can be made beginning 12 months after publication and for up to 36 months post publication. Deidentified individual participant data reported in the manuscript will be shared under the terms of a Data Use Agreement and may only be used for approved proposals. Requests may be made to: crdatashare@mskcc.org.

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/mskcc/html/44.cfm